CLINICAL TRIAL: NCT03695562
Title: Stability of Dental Implants Placed in Patients With Vitamin D Deficiency Using Sequential Drilling Versus a New One Single Drilling Design: A Randomized Clinical Trial
Brief Title: Stability of Dental Implants Placed in Patients With Vitamin D Deficiency Using Sequential Drilling Versus a New One Single Drilling Design
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Nabil Ahmed Younis, Teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: perio21005
Record Dates: First submitted 2018-09-30; First posted 2018-10-04 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Implant Stability With Vitamin D Deficiency
Keywords: vitamin D; implant stability; sequential drilling; single drilling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- implant placement using sequential drilling (Experimental): patient with vitamin D deficiency using sequential drilling technique
  Interventions: Procedure: sequential drilling technique
- implant placement using single drilling (Active Comparator): Patient with vitamin D deficiency using single drilling technique
  Interventions: Procedure: sequential drilling technique

INTERVENTIONS:
Procedure: sequential drilling technique — Patient with vitamin D deficiency using sequential drilling technique
  Other Names: conventional implant placement

SUMMARY:
- Vitamin D considers as the most potent effect on calcium level in blood it was found that vitamin D target mainly bone tissue intestine and kidney for calcium absorption In bone, vitamin D stimulates mainly the activity of osteoclasts osteoblast activity on the other hand it increases the production of extracellular matrix proteins by different osteoblastic activity. Vitamin D also increase intestinal calcium absorption and regulate synthesis and secretion of parathyroid hormone (PTH)

Implant consider as one of the most successful treatment modalities that usually used in dental clinics for restoring single or multiple missed teeth knowing that successful rate of dental implant may reach up to 99% however there are many different techniques for implant placement they mainly depend on the same procedure for implant placement even sequential drilling technique or single drilling technique some paper supported that sequential drilling is much better than single drilling technique on other hand some assume that single drilling is much better as it save time effort material less bone trauma & less heat generation although there are many studies performed on sequential drilling & single drilling techniques we still have a gap for understanding the ideal technique for implant placement in patients with vitamin D deficiency

DETAILED DESCRIPTION:
The high predictability of dental implants has led to routine use with a great expectation for success There are many researches focused on the outcome of delayed dental implant Since the first report of highly success rate after placement of a dental implant there has been increasing interest in this technique for implant treatment The goal of modern dentistry is to restore the patient's dentition to normal contour function comfort esthetics speech and health regardless of the atrophy disease or injury of the stomatognathic system As a result of disease related tooth loss and the value placed upon teeth there has been a continual search for methods by which missing teeth could be replaced Early artificial replacements were made from natural teeth and a variety of substitute materials All transplantation of a tooth from one person to another was an early method by which lost teeth were replaced Archeological discoveries indicate that many ancient civilizations practiced allogenic tooth transplantation. In 1561 Ambrose Pare reported that decayed teeth could be replaced by using extracted teeth from another individual and is credited with being the first to mention transplantation The core objective of dental implant therapy is to improve functional dentition throughout life Nevertheless there are many factors that may effect on implant stability A significant part of implant failure may be related to systemic condition that my retard dental implants osteointegration one of this factors is vitamin D deficiency recently many paper focused on vitamin D deficiency and its impact effect on bone turn over around dental implant There are many different techniques for implant placement even sequential drilling or single drilling technique knowing that single drilling technique has a compression effect which may enhance implant stability however sequential drilling don't have compression effect on bone some paper supported that sequential is much better than single drilling technique however some paper showed there is no clinical significance between two techniques the main idea here that we need to find an ideal technique for implant placement in patients with vitamin D deficiency knowing that vitamin D play an important role for bone turnover around dental implant to attain the required dental implant stability also play a role for osteoblast osteoclast activity Also vitamin D play a role for regulation of parathyroid hormone which play a role for homeostasis of calcium level from bone in blood .

ELIGIBILITY:
Inclusion criteria:

1. Age: 18-70.
2. Patient with vitamin D deficiency (< 30 ng/ml )
3. Patients with single or multiple missed teeth in upper & lower molar premolar area.
4. Patients with adequate bone volume for the dental implant procedure.
5. Patient with sufficient interarch space.
6. Patients who are compliant to oral hygiene measures.
7. Patient consent approval and signing.

Exclusion criteria:

1. Systemic disease that contraindicates implant placement or surgical procedures.
2. Poor patient's compliance.
3. Psychological problems.
4. Pathology at the site of intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2021-02-14 (Actual)

PRIMARY OUTCOMES:
primary/secondary implant stability | 6 months
  primary & secondary implant stability using ostell/periotest

SECONDARY OUTCOMES:
Swelling | 10 days
  post operative swelling questionnaire yes/no
post operative Pain: NRS | 10 days
  post operative pain by numerical rating scale from 0 to 10 , 0 no pain , 10 severe pain
bone resorption | 6 months
  crestal bone resorption :Digital radiography: Digora unit: mm

CONTACTS AND LOCATIONS:
Overall Officials: Amr zahran, Phd, Study Chair — Cairo University; Jehan Madkour, Phd, Study Chair — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
i will check with my supervisor

REFERENCES:
- [Result] Merheb J, Temmerman A, Rasmusson L, Kubler A, Thor A, Quirynen M. Influence of Skeletal and Local Bone Density on Dental Implant Stability in Patients with Osteoporosis. Clin Implant Dent Relat Res. 2016 Apr;18(2):253-60. doi: 10.1111/cid.12290. Epub 2016 Feb 10. PMID 26864614